CLINICAL TRIAL: NCT00033462
Title: A Phase II Trial of OSI-774 in Patients With Hepatocellular or Biliary Carcinoma
Brief Title: Erlotinib in Treating Patients With Unresectable Liver, Bile Duct, or Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02797; MC0152; 5429; N01CM17104 (NIH)
Record Dates: First submitted 2002-04-09; First posted 2003-06-06 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Primary Cholangiocellular Carcinoma; Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Erlotinib Hydrochloride

ARMS (1):
- Arm I (Experimental): Patients receive oral erlotinib once daily. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of erlotinib in treating patients who have unresectable liver, bile duct, or gallbladder cancer. Biological therapies such as erlotinib may interfere with the growth of cancer cells and slow the growth of the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the proportion of patients with unresectable hepatocellular or biliary carcinoma treated with OSI-774 who are progression-free at 24 weeks.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of this treatment in each of the patient groups.

II. To evaluate the objective response rate of patients with hepatocellular or biliary carcinoma treated with OSI-774.

III. To evaluate overall and progression-free survival. IV. To assess the EGFR protein levels and explore their association with clinical outcome.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 groups according to cancer type (hepatocellular vs biliary).

Patients receive oral erlotinib once daily. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC) or biliary carcinoma that is surgically unresectable; exception: for surgically unresectable HCC, a hypervascular mass on CT and an AFP > 100ng/mL will suffice as noninvasive diagnostic criteria
* Measurable disease defined as at least one lesion whose longest diameter can be accurately measured as ≥ 2.0 cm
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* PLT ≥ 75,000/mm3
* Total bilirubin ≤ 2 x upper normal limits (UNL)
* Serum AST ≤ 3 x UNL
* Serum ALT ≤ 3 x UNL
* Serum creatinine ≤ 2 mg/dL
* Serum albumin ≥ 2.5 g/dL
* Patients not receiving anticoagulation: INR ≤ 1.5
* ECOG performance status (PS) 0, 1, or 2
* Estimated life expectancy ≥ 3 months
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide written informed consent
* HCC Patients Only: Child-Pugh classification of A or B
* For patients having prior cryotherapy, radiofrequency ablation, ethanol injection, or photodynamic therapy, the following criteria must be met:

  * > 6 weeks has elapsed since that therapy
  * Indicator lesion(s) is/are outside the area of prior treatment or, if the only indicator lesion is inside the prior treatment area, there must be clear evidence of disease progression associated with that lesion
  * Edges of the indicator lesion are clearly distinct on CT scanning

Exclusion Criteria:

* Ampulla of Vater tumors
* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
  * NOTE: The effects of OSI-774 on the developing human fetus at the recommended therapeutic dose are unknown
* Any of the following:

  * > 1 prior systemic anticancer therapy; Note: Chemoembolization will be considered as one prior chemotherapeutic regimen.
  * Prior EGFR targeting therapy
  * Nitrosoureas or mitomycin C ≤6 weeks prior to study entry
  * Other chemotherapy ≤4 weeks prior to study entry

    • Immunotherapy ≤ 4 weeks prior to study entry
  * Biologic therapy ≤ 4 weeks prior to study entry
  * Radiation therapy ≤ 4 weeks prior to study entry
  * Prior cryotherapy, radiofrequency ablation, ethanol injection or photodynamic therapy ≤6 weeks prior to study entry
  * Failure to fully recover from adverse effects of prior therapies regardless of interval since last treatment
  * Other concurrent chemotherapy, immunotherapy, radiotherapy, or any other therapy or supportive care considered investigational
  * Major surgery, or significant traumatic injury occurring ≤ 3 weeks prior to planned treatment start date
* Any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior procedures affecting absorption
  * Active peptic ulcer disease
* History of other malignancy other than hepatocellular or biliary carcinoma within the previous 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma of the cervix
* Known abnormalities of the cornea such as:

  * History of dry eye syndrome or Sjorgen's syndrome
  * Congenital abnormality (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose)
  * Abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Known CNS metastases; NOTE: These patients are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy; NOTE: Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; these patients are excluded from the study because of possible pharmacokinetic interactions with OSI-774; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2002-03; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are progression-free at 24 weeks | At 24 weeks
  Confidence intervals for the true PFR will be calculated using the methods of Duffy-Santner.

SECONDARY OUTCOMES:
Objective response, defined by the RECIST criteria in terms of tumor/lesion size and change | Up to 3 years
Overall survival | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
EGFR protein levels | Baseline
  We will evaluate these EGFR protein levels and explore their association with clinical outcome.
Overall response rate in EGFR positive patients | Up to 3 years
  Analyses will be done independently on patients from each patient group. Corresponding 95% confidence intervals will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Philip, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States